CLINICAL TRIAL: NCT03095105
Title: An Open-label, Parallel-group Study to Compare the Pharmacokinetic Profile in Healthy Elderly Subjects Versus Healthy Young Subjects After Single and Repeated Oral Administration of BIA 6-512 (Trans-resveratrol)
Brief Title: Pharmacokinetic Profile of BIA 6-512 in Healthy Elderly Subjects Versus Healthy Young Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-6512-105
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young group (Experimental): The study was performed in two consecutive phases: single-dose and multiple-dose.
  Subjects were institutionalised on Day 0, the day prior to the single-dose administration (Day 1). Single dose (dose 1) of BIA 6-512 200 mg was administered on Day 1 and subjects remained confined in the Unit until the 24 h post-dose procedures (Day 2). Then, subjects started being administered BIA 6-512 200 mg thrice-daily until the morning of Day 4 (Dose 8). Blood samples were taken at pre-determined time-points for the assay of BIA 6-512
  Interventions: Drug: 200 mg BIA 6-512
- Elderly group (Experimental): The study was performed in two consecutive phases: single-dose and multiple-dose.
  Subjects were institutionalised on Day 0, the day prior to the single-dose administration (Day 1). Single dose (dose 1) of BIA 6-512 200 mg was administered on Day 1 and subjects remained confined in the Unit until the 24 h post-dose procedures (Day 2). Then, subjects started being administered BIA 6-512 200 mg thrice-daily until the morning of Day 4 (Dose 8). Blood samples were taken at pre-determined time-points for the assay of BIA 6-512
  Interventions: Drug: 200 mg BIA 6-512

INTERVENTIONS:
Drug: 200 mg BIA 6-512 — capsules containing BIA 6-512 200 mg was administered orally, with 240 mL of mineral water without gas at room tempera¬ture
  Other Names: Trans-resveratrol

SUMMARY:
the purpose of the study was to the compare pharmacokinetic profile of BIA 6-512 in healthy elderly subjects versus healthy young subjects after single and repeated oral administration of 200 mg BIA 6-512.

DETAILED DESCRIPTION:
Single-centre, open-label study in healthy young (18-40 years) and elderly (65 years or older) subjects. The study consisted of a single-dose phase followed by a repeated dose phase (3 times daily, at 8-h intervals). Subjects were admitted on the day prior to the first dose (Day 1). On day 1, a single dose of 200 mg BIA 6-512 (Dose 1) was administered in the morning. On day 2, the repeated dose phase started 24 h post first dosing. In the repeated dose phase (Doses 2 to 8) subjects received 200 mg BIA 6-512 every 8 hours until the morning of day 4 (approximately 72 hours post first dosing).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 40 years, inclusive (young); or male or female subjects aged 65 years or more (elderly).
* Body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Healthy as determined by an inter¬view, pre-study medical history, physical examination, vital signs, neurological examination and 12-lead ECG; clinical laboratory test results clinically acceptable at screening and admission.
* Negative tests for HBsAg, anti-HCVAb, anti-HIV-1 Ab and anti-HIV-2 Ab at screening.
* Negative screen for drugs of abuse at screening and admission.
* Informed consent signed by the subject.
* Co-operative and available for the entire study.
* Abstinence from alcohol for 48 hours prior to admission (as stated by subject). An alcohol breath test performed at screening and at admission to the clinic had to be negative.
* Non-smokers or who smoke ≤ 10 cigarettes or equivalent per day.
* If female, in the young group: She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence; and she had a negative urine pregnancy test at screening and admission.

Exclusion Criteria:

* Evidence in the subject's medical history or in the medical exa¬mina¬tion of any clinically significant respiratory, hepatic, renal, gastrointesti¬nal, haematological, lymphatic, neurological, car¬diovascu¬lar, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue or other significant acute or chronic abnormalities which might influence either the safety of the subject or the ab¬sorption, dis¬tribution, meta¬bolism or excretion of the active agent under investigation.
* History of relevant drug or food hypersensitivity.
* Significant infection or known inflammatory process on screening or admission.
* Acute gastrointestinal symptoms at the time of screening or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Regular use of any medication within four weeks prior to study admission (self-medication or prescription).
* Single use of any medication (including OTC) that was not expressly permitted within two weeks prior admission to the stu¬dy.
* Abuse of alcohol (equiv¬alent to more than 35 g ethanol per day).
* Vegetarians, vegans or subjects who had medical dietary restrictions.
* History of alcoholism or drug abuse.
* Participation in a clinical investigation within two months prior to screening.
* Blood donation of more than 250 ml within two months prior to screening. Blood donation of less than 250 ml or plasma donation with¬in one month prior to screening.
* Subjects who were known or suspected:

  * not to comply with the study directives
  * not to be reliable or trustworthy
  * not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed
  * to be in such a precarious financial situation that they no longer weigh up the possible risks of their participation and the unpleasantness they may be involved in.
* If female, in the young group: she was pregnant or breast-feeding; she was of childbearing potential and she did not use an approved effective contraceptive method (double-barrier, intra-uterine device or abstinence) or she used oral contraceptives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-01-24 (Actual); Primary Completion 2006-03-02 (Actual); Study Completion 2006-03-02 (Actual)

PRIMARY OUTCOMES:
Cmax - the maximum observed plasma concentration (single dose) | Day 1: pre-dose 1, and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12 and 16 h post-dose
AUCτ- the area under the plasma concentration versus time curve over the dosing interval, calculated by the linear trapezoidal rule (Single dose) | Day 1: pre-dose 1, and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12 and 16 h post-dose
AUC0-∞ - the area under the plasma concentration versus time curve from time zero to infinity, calculated from AUC0-t + (Clast/lz ), where Clast is the last quantifiable concentration. (single dose) | Day 1: pre-dose 1, and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12 and 16 h post-dose
Cmax - the maximum observed plasma concentration (multiple dose) | Day 2: pre-dose 2; pre-dose 3 and pre-dose 4; day 3: pre-dose 5, pre-dose 6 and pre-dose 7; day 4: pre-dose 8 and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12 and 16 h post-dose; day 5: 24 h after last dose (dose 8).
  Effect of age on the BIA 6-512 pharmacokinetics
AUCτ - the area under the plasma concentration versus time curve over the dosing interval, calculated by the linear trapezoidal rule (multiple dose) | Day 2: pre-dose 2; pre-dose 3 and pre-dose 4; day 3: pre-dose 5, pre-dose 6 and pre-dose 7; day 4: pre-dose 8 and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12 and 16 h post-dose; day 5: 24 h after last dose (dose 8).
  Effect of age on the BIA 6-512 pharmacokinetics
AUC0-∞ - the area under the plasma concentration versus time curve from time zero to infinity, calculated from AUC0-t + (Clast/lz ), where Clast is the last quantifiable concentration. (multiple dose) | Day 2: pre-dose 2; pre-dose 3 and pre-dose 4; day 3: pre-dose 5, pre-dose 6 and pre-dose 7; day 4: pre-dose 8 and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12 and 16 h post-dose; day 5: 24 h after last dose (dose 8).
  Effect of age on the BIA 6-512 pharmacokinetics

CONTACTS AND LOCATIONS:
Locations (1):
- Scope International AG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided